CLINICAL TRIAL: NCT00272428
Title: The SU.VI.MAX Study. A Randomized, Placebo-controlled Prevention Trial of the Health Effects of Antioxidant Vitamins and Minerals.
Brief Title: Primary Prevention Trial of the Health Effects of Antioxidant Vitamins and Minerals.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: French private agencies (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 94-706
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2007-10

CONDITIONS: Healthy
Keywords: Prevention trial; Antioxydant vitamins and minerals; Cancer; Ischemic disease; Mortality; Health related quality of life
MeSH Terms: conditions — Neoplasms | interventions — Ascorbic Acid; Vitamin E; beta Carotene; Selenium; Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: ascorbic acid, vitamin E, beta carotene, selenium, zinc

SUMMARY:
It has been suggested that a low dietary intake of antioxidant vitamins and minerals increases the incidence rate of cardiovascular disease and cancer. To date, however, the published results of randomized, placebo-controlled trials of supplements containing antioxidant nutrients have not provided clear evidence of a beneficial effect. We tested the efficacy of nutritional doses of supplementation with a combination of antioxidant vitamins and minerals in reducing the incidence of cancer and ischemic cardiovascular disease in the general population.

DETAILED DESCRIPTION:
From experimental studies it is known that free radicals may induce numerous pathological processes, and it has been suggested that, because of their antioxidant capacity, nutrients such as beta-carotene, vitamin C, vitamin E, selenium and zinc may prevent such harmful effects. Epidemiological data from cross-sectional, case-control, and prospective studies have indeed shown a strong relationship between the intake of antioxidant vitamins and minerals, or foods rich in these nutrients, and the risk of cancer and ischaemic cardiovascular diseases (CVD). However, randomised placebo-controlled primary prevention trials, in which antioxidant micronutrients alone or in pairs were given at high doses over long periods, have not been able to prove this potential beneficial effect, and two of these even suggested harmful effects. The seemingly contradictory results between the observational studies and these randomised trials can be explained by the fact that the doses used in clinical trials were much higher than the highest levels reachable by usual dietary intake which have been found to be associated in observational studies with the lowest risk of cancer and CVD. In fact, the only trial which did observe a beneficial effect on total mortality and cancer incidence used nutritional doses of a combination of several vitamins and minerals and was performed on Chinese population with very low baseline micronutrient status, due to poor life conditions in this region (9).

The objective of the "SUpplementation en VItamines et Minéraux AntioXydants" (SU.VI.MAX) study, was to test in a randomised, placebo-controlled trial, if an adequate and well balanced intake of antioxidant nutrients reduces the incidence of cancers and ischaemic cardiovascular diseases in a middle-age general population.

ELIGIBILITY:
Inclusion Criteria:

* women aged 35-60 years, men aged 45-60 years
* acceptance of the possibility to be given a placebo and acceptance of the constraints of participation
* lack of previous regular supplementation with any of the vitamins or minerals in the supplement provided
* absence of extreme beliefs or behavior regarding diet

Exclusion Criteria:

* disease likely to hinder active participation or threatened 5-year survival

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13000
Dates: Start 1994-10; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Major fatal and non fatal ischemic cardiovascular events
Cancer any kind except for basal cell skin carcinoma

SECONDARY OUTCOMES:
All cause mortality
Health-related quality of life
Intermediate criteria of clinical status
Intermediate criteria of biological status
Intermediate criteria of anthropometric status

CONTACTS AND LOCATIONS:
Overall Officials: Serge Hercberg, MD, PhD, Principal Investigator — U557 Inserm (UMR Inserm/Inra/CNAM), Institut Scientifique et Technique de la Nutrition et de l'Alimentation/CNAM
Locations (1):
- U557 Inserm, Paris, France

REFERENCES:
- [Result] Hercberg S, Galan P, Preziosi P, Bertrais S, Mennen L, Malvy D, Roussel AM, Favier A, Briancon S. The SU.VI.MAX Study: a randomized, placebo-controlled trial of the health effects of antioxidant vitamins and minerals. Arch Intern Med. 2004 Nov 22;164(21):2335-42. doi: 10.1001/archinte.164.21.2335. PMID 15557412
- [Derived] Andreeva VA, Peneau S, Julia C, Shivappa N, Hebert JR, Wirth MD, Touvier M, Hercberg S, Galan P, Kesse-Guyot E. The inflammatory potential of the diet is prospectively associated with subjective hearing loss. Eur J Nutr. 2021 Oct;60(7):3669-3678. doi: 10.1007/s00394-021-02531-1. Epub 2021 Mar 18. PMID 33738534
- [Derived] Lecuyer L, Dalle C, Micheau P, Petera M, Centeno D, Lyan B, Lagree M, Galan P, Hercberg S, Rossary A, Demidem A, Vasson MP, Partula V, Deschasaux M, Srour B, Latino-Martel P, Druesne-Pecollo N, Kesse-Guyot E, Durand S, Pujos-Guillot E, Manach C, Touvier M. Untargeted plasma metabolomic profiles associated with overall diet in women from the SU.VI.MAX cohort. Eur J Nutr. 2020 Dec;59(8):3425-3439. doi: 10.1007/s00394-020-02177-5. Epub 2020 Jan 11. PMID 31927670
- [Derived] Lecuyer L, Dalle C, Lyan B, Demidem A, Rossary A, Vasson MP, Petera M, Lagree M, Ferreira T, Centeno D, Galan P, Hercberg S, Deschasaux M, Partula V, Srour B, Latino-Martel P, Kesse-Guyot E, Druesne-Pecollo N, Durand S, Pujos-Guillot E, Touvier M. Plasma Metabolomic Signatures Associated with Long-term Breast Cancer Risk in the SU.VI.MAX Prospective Cohort. Cancer Epidemiol Biomarkers Prev. 2019 Aug;28(8):1300-1307. doi: 10.1158/1055-9965.EPI-19-0154. Epub 2019 Jun 4. PMID 31164347
- [Derived] Assmann KE, Adjibade M, Hercberg S, Galan P, Kesse-Guyot E. Unsaturated Fatty Acid Intakes During Midlife Are Positively Associated with Later Cognitive Function in Older Adults with Modulating Effects of Antioxidant Supplementation. J Nutr. 2018 Dec 1;148(12):1938-1945. doi: 10.1093/jn/nxy206. PMID 30517725
- [Derived] Wiernik E, Lemogne C, Fezeu L, Arnault N, Hercberg S, Kesse-Guyot E, Galan P. Association Between Alexithymia and Risk of Incident Cardiovascular Diseases in the SUpplementation en VItamines et Mineraux AntioXydants (SU.VI.MAX) Cohort. Psychosom Med. 2018 Jun;80(5):460-467. doi: 10.1097/PSY.0000000000000592. PMID 29649036
- [Derived] Assmann KE, Adjibade M, Shivappa N, Hebert JR, Wirth MD, Touvier M, Akbaraly T, Hercberg S, Galan P, Julia C, Kesse-Guyot E. The Inflammatory Potential of the Diet at Midlife Is Associated with Later Healthy Aging in French Adults. J Nutr. 2018 Mar 1;148(3):437-444. doi: 10.1093/jn/nxx061. PMID 29546305
- [Derived] Ruhunuhewa I, Adjibade M, Andreeva VA, Galan P, Hercberg S, Assmann KE, Kesse-Guyot E. Prospective association between body mass index at midlife and healthy aging among French adults. Obesity (Silver Spring). 2017 Jul;25(7):1254-1262. doi: 10.1002/oby.21853. Epub 2017 May 11. PMID 28494135
- [Derived] Adjibade M, Andreeva VA, Lemogne C, Touvier M, Shivappa N, Hebert JR, Wirth MD, Hercberg S, Galan P, Julia C, Assmann KE, Kesse-Guyot E. The Inflammatory Potential of the Diet Is Associated with Depressive Symptoms in Different Subgroups of the General Population. J Nutr. 2017 May;147(5):879-887. doi: 10.3945/jn.116.245167. Epub 2017 Mar 29. PMID 28356432
- [Derived] Walker V, Perret-Guillaume C, Kesse-Guyot E, Agrinier N, Hercberg S, Galan P, Assmann KE, Briancon S, Rotonda C. Effect of Multimorbidity on Health-Related Quality of Life in Adults Aged 55 Years or Older: Results from the SU.VI.MAX 2 Cohort. PLoS One. 2016 Dec 29;11(12):e0169282. doi: 10.1371/journal.pone.0169282. eCollection 2016. PMID 28033414
- [Derived] Kesse-Guyot E, Assmann KE, Andreeva VA, Touvier M, Neufcourt L, Shivappa N, Hebert JR, Wirth MD, Hercberg S, Galan P, Julia C. Long-term association between the dietary inflammatory index and cognitive functioning: findings from the SU.VI.MAX study. Eur J Nutr. 2017 Jun;56(4):1647-1655. doi: 10.1007/s00394-016-1211-3. Epub 2016 Apr 7. PMID 27055851
- [Derived] Adriouch S, Julia C, Kesse-Guyot E, Mejean C, Ducrot P, Peneau S, Donnenfeld M, Deschasaux M, Menai M, Hercberg S, Touvier M, Fezeu LK. Prospective association between a dietary quality index based on a nutrient profiling system and cardiovascular disease risk. Eur J Prev Cardiol. 2016 Oct;23(15):1669-76. doi: 10.1177/2047487316640659. Epub 2016 Mar 21. PMID 27000099
- [Derived] Graffouillere L, Deschasaux M, Mariotti F, Neufcourt L, Shivappa N, Hebert JR, Wirth MD, Latino-Martel P, Hercberg S, Galan P, Julia C, Kesse-Guyot E, Touvier M. The Dietary Inflammatory Index Is Associated with Prostate Cancer Risk in French Middle-Aged Adults in a Prospective Study. J Nutr. 2016 Apr 1;146(4):785-791. doi: 10.3945/jn.115.225623. Epub 2016 Mar 9. PMID 26962176
- [Derived] Graffouillere L, Deschasaux M, Mariotti F, Neufcourt L, Shivappa N, Hebert JR, Wirth MD, Latino-Martel P, Hercberg S, Galan P, Julia C, Kesse-Guyot E, Touvier M. Prospective association between the Dietary Inflammatory Index and mortality: modulation by antioxidant supplementation in the SU.VI.MAX randomized controlled trial. Am J Clin Nutr. 2016 Mar;103(3):878-85. doi: 10.3945/ajcn.115.126243. Epub 2016 Feb 10. PMID 26864363
- [Derived] Deschasaux M, Souberbielle JC, Latino-Martel P, Sutton A, Charnaux N, Druesne-Pecollo N, Galan P, Hercberg S, Le Clerc S, Kesse-Guyot E, Ezzedine K, Touvier M. Weight Status and Alcohol Intake Modify the Association between Vitamin D and Breast Cancer Risk. J Nutr. 2016 Mar;146(3):576-85. doi: 10.3945/jn.115.221481. Epub 2016 Jan 27. PMID 26817718
- [Derived] Kesse-Guyot E, Assmann KE, Andreeva VA, Ferry M, Hercberg S, Galan P; SU.VI.MAX 2 Research Group. Consumption of Dairy Products and Cognitive Functioning: Findings from the SU.VI.MAX 2 Study. J Nutr Health Aging. 2016 Feb;20(2):128-37. doi: 10.1007/s12603-015-0593-x. PMID 26812508
- [Derived] Deschasaux M, Souberbielle JC, Latino-Martel P, Sutton A, Charnaux N, Druesne-Pecollo N, Galan P, Hercberg S, Le Clerc S, Kesse-Guyot E, Ezzedine K, Touvier M. Prospective associations between vitamin D status, vitamin D-related gene polymorphisms, and risk of tobacco-related cancers. Am J Clin Nutr. 2015 Nov;102(5):1207-15. doi: 10.3945/ajcn.115.110510. Epub 2015 Oct 7. PMID 26447153
- [Derived] Kesse-Guyot E, Lassale C, Assmann KE, Andreeva VA, Julia C, Blacher J, Fezeu L, Hercberg S, Galan P. Are different vascular risk scores calculated at midlife uniformly associated with subsequent poor cognitive performance? Atherosclerosis. 2015 Nov;243(1):286-92. doi: 10.1016/j.atherosclerosis.2015.09.023. Epub 2015 Sep 21. PMID 26409628
- [Derived] Donnenfeld M, Deschasaux M, Latino-Martel P, Diallo A, Galan P, Hercberg S, Ezzedine K, Touvier M. Prospective association between dietary folate intake and skin cancer risk: results from the Supplementation en Vitamines et Mineraux Antioxydants cohort. Am J Clin Nutr. 2015 Aug;102(2):471-8. doi: 10.3945/ajcn.115.109041. Epub 2015 Jul 8. PMID 26156743
- [Derived] Chhim AS, Fassier P, Latino-Martel P, Druesne-Pecollo N, Zelek L, Duverger L, Hercberg S, Galan P, Deschasaux M, Touvier M. Prospective association between alcohol intake and hormone-dependent cancer risk: modulation by dietary fiber intake. Am J Clin Nutr. 2015 Jul;102(1):182-9. doi: 10.3945/ajcn.114.098418. Epub 2015 May 20. PMID 25994566
- [Derived] Kesse-Guyot E, Andreeva VA, Touvier M, Jeandel C, Ferry M, Hercberg S, Galan P; SU.VI.MAX 2 Research Group. Overall and abdominal adiposity in midlife and subsequent cognitive function. J Nutr Health Aging. 2015 Feb;19(2):183-9. doi: 10.1007/s12603-014-0508-2. PMID 25651444
- [Derived] Deschasaux M, Pouchieu C, His M, Hercberg S, Latino-Martel P, Touvier M. Dietary total and insoluble fiber intakes are inversely associated with prostate cancer risk. J Nutr. 2014 Apr;144(4):504-10. doi: 10.3945/jn.113.189670. Epub 2014 Feb 19. PMID 24553693
- [Derived] Touvier M, Deschasaux M, Montourcy M, Sutton A, Charnaux N, Kesse-Guyot E, Fezeu LK, Latino-Martel P, Druesne-Pecollo N, Malvy D, Galan P, Hercberg S, Ezzedine K, Souberbielle JC. Interpretation of plasma PTH concentrations according to 25OHD status, gender, age, weight status, and calcium intake: importance of the reference values. J Clin Endocrinol Metab. 2014 Apr;99(4):1196-203. doi: 10.1210/jc.2013-3349. Epub 2014 Feb 14. PMID 24527713
- [Derived] Andreeva VA, Galan P, Arnaud J, Julia C, Hercberg S, Kesse-Guyot E. Midlife iron status is inversely associated with subsequent cognitive performance, particularly in perimenopausal women. J Nutr. 2013 Dec;143(12):1974-81. doi: 10.3945/jn.113.177089. Epub 2013 Oct 2. PMID 24089418
- [Derived] Julia C, Touvier M, Meunier N, Papet I, Galan P, Hercberg S, Kesse-Guyot E. Intakes of PUFAs were inversely associated with plasma C-reactive protein 12 years later in a middle-aged population with vitamin E intake as an effect modifier. J Nutr. 2013 Nov;143(11):1760-6. doi: 10.3945/jn.113.180943. Epub 2013 Sep 11. PMID 24027184
- [Derived] Kesse-Guyot E, Andreeva VA, Jeandel C, Ferry M, Touvier M, Hercberg S, Galan P. Alcohol consumption in midlife and cognitive performance assessed 13 years later in the SU.VI.MAX 2 cohort. PLoS One. 2012;7(12):e52311. doi: 10.1371/journal.pone.0052311. Epub 2012 Dec 19. PMID 23284983
- [Derived] Kesse-Guyot E, Andreeva VA, Lassale C, Ferry M, Jeandel C, Hercberg S, Galan P; SU.VI.MAX 2 Research Group. Mediterranean diet and cognitive function: a French study. Am J Clin Nutr. 2013 Feb;97(2):369-76. doi: 10.3945/ajcn.112.047993. Epub 2013 Jan 2. PMID 23283500
- [Derived] Kesse-Guyot E, Charreire H, Andreeva VA, Touvier M, Hercberg S, Galan P, Oppert JM. Cross-sectional and longitudinal associations of different sedentary behaviors with cognitive performance in older adults. PLoS One. 2012;7(10):e47831. doi: 10.1371/journal.pone.0047831. Epub 2012 Oct 17. PMID 23082222
- [Derived] Kesse-Guyot E, Ahluwalia N, Lassale C, Hercberg S, Fezeu L, Lairon D. Adherence to Mediterranean diet reduces the risk of metabolic syndrome: a 6-year prospective study. Nutr Metab Cardiovasc Dis. 2013 Jul;23(7):677-83. doi: 10.1016/j.numecd.2012.02.005. Epub 2012 May 25. PMID 22633793
- [Derived] Touvier M, Kesse-Guyot E, Andreeva VA, Fezeu L, Charnaux N, Sutton A, Druesne-Pecollo N, Hercberg S, Galan P, Zelek L, Latino-Martel P, Czernichow S. Modulation of the association between plasma intercellular adhesion molecule-1 and cancer risk by n-3 PUFA intake: a nested case-control study. Am J Clin Nutr. 2012 Apr;95(4):944-50. doi: 10.3945/ajcn.111.027805. Epub 2012 Feb 29. PMID 22378736
- [Derived] Briancon S, Boini S, Bertrais S, Guillemin F, Galan P, Hercberg S. Long-term antioxidant supplementation has no effect on health-related quality of life: the randomized, double-blind, placebo-controlled, primary prevention SU.VI.MAX trial. Int J Epidemiol. 2011 Dec;40(6):1605-16. doi: 10.1093/ije/dyr161. PMID 22158670
- [Derived] Peneau S, Galan P, Jeandel C, Ferry M, Andreeva V, Hercberg S, Kesse-Guyot E; SU.VI.MAX 2 Research Group. Fruit and vegetable intake and cognitive function in the SU.VI.MAX 2 prospective study. Am J Clin Nutr. 2011 Nov;94(5):1295-303. doi: 10.3945/ajcn.111.014712. Epub 2011 Sep 28. PMID 21955649
- [Derived] Kesse-Guyot E, Fezeu L, Jeandel C, Ferry M, Andreeva V, Amieva H, Hercberg S, Galan P. French adults' cognitive performance after daily supplementation with antioxidant vitamins and minerals at nutritional doses: a post hoc analysis of the Supplementation in Vitamins and Mineral Antioxidants (SU.VI.MAX) trial. Am J Clin Nutr. 2011 Sep;94(3):892-9. doi: 10.3945/ajcn.110.007815. Epub 2011 Jul 20. PMID 21775560
- [Derived] Perez-Jimenez J, Fezeu L, Touvier M, Arnault N, Manach C, Hercberg S, Galan P, Scalbert A. Dietary intake of 337 polyphenols in French adults. Am J Clin Nutr. 2011 Jun;93(6):1220-8. doi: 10.3945/ajcn.110.007096. Epub 2011 Apr 13. PMID 21490142
- [Derived] Kesse-Guyot E, Amieva H, Castetbon K, Henegar A, Ferry M, Jeandel C, Hercberg S, Galan P; SU.VI.MAX 2 Research Group. Adherence to nutritional recommendations and subsequent cognitive performance: findings from the prospective Supplementation with Antioxidant Vitamins and Minerals 2 (SU.VI.MAX 2) study. Am J Clin Nutr. 2011 Jan;93(1):200-10. doi: 10.3945/ajcn.2010.29761. Epub 2010 Nov 24. PMID 21106918
- [Derived] Ezzedine K, Latreille J, Kesse-Guyot E, Galan P, Hercberg S, Guinot C, Malvy D. Incidence of skin cancers during 5-year follow-up after stopping antioxidant vitamins and mineral supplementation. Eur J Cancer. 2010 Dec;46(18):3316-22. doi: 10.1016/j.ejca.2010.06.008. Epub 2010 Jul 6. PMID 20605091
- [Derived] Kesse-Guyot E, Vergnaud AC, Fezeu L, Zureik M, Blacher J, Peneau S, Hercberg S, Galan P, Czernichow S. Associations between dietary patterns and arterial stiffness, carotid artery intima-media thickness and atherosclerosis. Eur J Cardiovasc Prev Rehabil. 2010 Dec;17(6):718-24. doi: 10.1097/HJR.0b013e32833a197f. PMID 20431391
- [Derived] Phillips CM, Goumidi L, Bertrais S, Field MR, Cupples LA, Ordovas JM, Defoort C, Lovegrove JA, Drevon CA, Gibney MJ, Blaak EE, Kiec-Wilk B, Karlstrom B, Lopez-Miranda J, McManus R, Hercberg S, Lairon D, Planells R, Roche HM. Gene-nutrient interactions with dietary fat modulate the association between genetic variation of the ACSL1 gene and metabolic syndrome. J Lipid Res. 2010 Jul;51(7):1793-800. doi: 10.1194/jlr.M003046. Epub 2010 Feb 22. PMID 20176858
- [Derived] Phillips CM, Goumidi L, Bertrais S, Ferguson JF, Field MR, Kelly ED, Peloso GM, Cupples LA, Shen J, Ordovas JM, McManus R, Hercberg S, Portugal H, Lairon D, Planells R, Roche HM. Complement component 3 polymorphisms interact with polyunsaturated fatty acids to modulate risk of metabolic syndrome. Am J Clin Nutr. 2009 Dec;90(6):1665-73. doi: 10.3945/ajcn.2009.28101. Epub 2009 Oct 14. PMID 19828715
- [Derived] Czernichow S, Vergnaud AC, Galan P, Arnaud J, Favier A, Faure H, Huxley R, Hercberg S, Ahluwalia N. Effects of long-term antioxidant supplementation and association of serum antioxidant concentrations with risk of metabolic syndrome in adults. Am J Clin Nutr. 2009 Aug;90(2):329-35. doi: 10.3945/ajcn.2009.27635. Epub 2009 Jun 2. PMID 19491388
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/16923246?ordinalpos=60&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum